CLINICAL TRIAL: NCT06045390
Title: Assessing the Effects of an In-office, Language-concordant App on Eye Drop Recall in Patients With Multi-drop Regimens
Brief Title: An App-based Instructional Platform to Improve Eye Drop Recall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-39908
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App arm (Experimental): The intervention is an in-office app that contains graphical and narrated information on a patient's specific drop regimen, and includes a quiz and a graphical print-out of their drop schedule. The patient will use the app during their clinic visit.
  Interventions: Other: App
- Standard arm (No Intervention): The standard arm will be the standard of care, which involves a provider explanation of their drop regimen (using a phone interpreter if needed).

INTERVENTIONS:
Other: App — App features (App will be used during the office visit):
  * Pictorial representation of drops (color-coded) and schedule.
  * Quiz to assess understanding of the regimen.
  * Narrated instructions (language-concordant) on how and when (frequency and eye laterality) to take each drop.
  * Graphical print-out of the regimen.
  Other Names: App-based drop instructions
  Arms: App arm

SUMMARY:
The goal of this interventional study is to assess whether an in-office, language-concordant instructional app improves drop regimen recall in a population of glaucoma patients who are on multi-drop regimens.

Participants will be divided into two groups -- those who use the app and those who do not. The app will have narrated information regarding the drop regimen, a quiz to test understanding of the regimen, and will enable a graphical printout of the eye drops and schedule.

At one month, both groups will be assessed on their eye drop regimen recall.

DETAILED DESCRIPTION:
Specific Aim: To investigate whether a language-concordant instructional application improves drop regimen recall in population of glaucoma patients at a 1-month follow-up period.

App features

1. Pictorial representation of drops (color-coded) and schedule.
2. Quiz to assess understanding of the regimen.
3. Narrated instructions (language-concordant) on how and when (frequency and eye laterality) to take each drop.
4. Graphical print-out of the regimen.

Study design

1. Study design: Randomized study, two groups: (1) patients that use the app, and (2) patients that do not use the app.
2. Study population:

   Inclusion criteria: patients with primary open-angle glaucoma on at least 2 eye drops

   Exclusion criteria: patients taking additional prescribed eye drops for other eye conditions; patients diagnosed within the last 3 months; patients unable to self-administer eye drops
3. Intervention: Use of an in-office app that has both graphical and verbal (language-concordant) instruction for how to use drops.
4. Main outcome measure: Ability to correctly identify drops/regimen

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of glaucoma (any type)
* drop regimen of at least 2 pressure-lowering drops
* languages supported at this time: English, Spanish, Cantonese

Exclusion Criteria:

* concurrent eye conditions necessitating additional eye drops
* inability to self-administer eye drops
* inability to engage with app (either visual or other barrier)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage accuracy of drop regimen recall | 1 month follow up from time of intervention
  This will be assessed through questions querying which drops the patients are taking, the number of times they are taking each drop, and the laterality of each drop. Each answer/drop will be individual recorded, and then total number of correct answers will be divided by the total number of questions.

SECONDARY OUTCOMES:
Overall medication adherence, assessed through the modified Morisky Adherence Scale, a widely published scale for general medication adherence | 1 month follow up from time of intervention
  An 8 question survey (7 questions are yes/no, with the final question on a Likert scale) gauging overall medication adherence. Each question will be individually assessed (not summed into a cumulative score). The higher number of "yes" responses corresponds to a lower adherence score.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Brodie, MD, Principal Investigator — UCSF, Department of Ophthalmology
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newman-Casey PA, Blachley T, Lee PP, Heisler M, Farris KB, Stein JD. Patterns of Glaucoma Medication Adherence over Four Years of Follow-Up. Ophthalmology. 2015 Oct;122(10):2010-21. doi: 10.1016/j.ophtha.2015.06.039. Epub 2015 Aug 25. PMID 26319441
- [Background] Zolnierek KB, Dimatteo MR. Physician communication and patient adherence to treatment: a meta-analysis. Med Care. 2009 Aug;47(8):826-34. doi: 10.1097/MLR.0b013e31819a5acc. PMID 19584762
- [Background] Newman-Casey PA, Robin AL, Blachley T, Farris K, Heisler M, Resnicow K, Lee PP. The Most Common Barriers to Glaucoma Medication Adherence: A Cross-Sectional Survey. Ophthalmology. 2015 Jul;122(7):1308-16. doi: 10.1016/j.ophtha.2015.03.026. Epub 2015 Apr 24. PMID 25912144